CLINICAL TRIAL: NCT03312543
Title: A Randomized, Evaluator-Blinded Clinical Study to Evaluate the Efficacy and Tolerability of an Investigational Light Therapy Mask on Subjects With Mild to Moderate Mottled Hyperpigmentation and Moderate to Severe Facial Wrinkles
Brief Title: Evaluation of the Efficacy and Tolerance of a Light Therapy Mask on Mild to Moderate Brown Spots and Moderate to Severe Facial Wrinkles
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Consumer Inc. (J&JCI) (Industry)
Responsible Party: Sponsor
Organization: Johnson & Johnson Consumer and Personal Products Worldwide (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CO-170511132943-SACT
Record Dates: First submitted 2017-10-06; First posted 2017-10-17 (Actual); Results first posted 2019-03-05 (Actual); Last update posted 2019-03-05 (Actual); Status verified 2019-02

CONDITIONS: Skin Aging
Keywords: Photoaging of Skin, Skin Wrinkling, Solar Aging of Skin, light therapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Active Cell: Active Mask (Experimental): Cleanser, Moisturizer, Active Mask
  Interventions: Device: Active Mask
- Sham Cell: Sham Mask (Sham Comparator): Cleanser, Moisturizer, Sham Mask
  Interventions: Device: Sham Mask

INTERVENTIONS:
Device: Active Mask — A facial cleanser will be used twice daily (morning and evening). In the morning after washing, the moisturizer with SPF will be applied full-face. For the first 12 weeks of the study, the active light therapy mask will be used for 10 minutes in the evening after washing/drying the face. For the second 12 weeks of the study, mask usage will be discontinued.
  Other Names: Active Light Therapy Mask
  Arms: Active Cell: Active Mask
Device: Sham Mask — A facial cleanser will be used twice daily (morning and evening). In the morning after washing, the moisturizer with SPF will be applied full-face. For the first 12 weeks of the study, the sham light therapy mask will be used for 10 minutes in the evening after washing/drying the face. For the second 12 weeks of the study, mask usage will be discontinued.
  Other Names: Sham Light Therapy Mask
  Arms: Sham Cell: Sham Mask

SUMMARY:
This research study will test how well a light therapy mask works for women with mild to moderate hyperpigmentation (brown spots) and moderate to severe facial wrinkles, as compared to a "sham" or inactive investigational light therapy mask. The study will also test if the light therapy mask causes any irritation. For the first 12 weeks of the study, participants will use the assigned mask, along with a provided cleanser and sunscreen. For the second 12 weeks of the study, participants will use just the cleanser and sunscreen.

DETAILED DESCRIPTION:
Exposure to sunlight and artificial light sources containing ultraviolet (UV) radiation is known to accelerate the skin's aging process, resulting in unwanted wrinkles, irregular skin tone, and loss of elasticity. Ablative techniques, such as dermabrasion, deep chemical peels, and ablative laser resurfacing of various wavelengths, are well documented to alleviate the signs of photodamage. However, such techniques often require significant post-treatment care and have higher risk profiles than other treatments, with potential side effects including erythema, pigmentation issues, infection, and possible scarring. They may be poorly tolerated by patients who dislike the discomfort, wound care, and prolonged downtime involved.

Non-ablative skin rejuvenation procedures are also effective for improving the appearance of photodamaged skin and are becoming increasingly popular because of their minimal downtime and increased safety. These procedures include intense pulsed light systems, non-ablative lasers, and monochromatic light boxes, which can target facial rhytids, irregular pigmentation, telangiectasia, and skin laxity. Unfortunately, such techniques can be expensive and their use is primarily limited to clinical settings.

However, the light-emitting diode (LED) is a novel light source that is well-suited for non-ablative phototherapy that can be utilized at home for a relatively low price. This study will evaluate the efficacy and tolerance of an LED-based light therapy mask as compared to a sham mask in subjects seeking anti-aging benefits.

ELIGIBILITY:
Inclusion Criteria:

* Has mild to moderate brown spots
* Has moderate to severe facial wrinkling
* Able to read, write, speak, and understand English
* In general good health
* If capable of having a child: must agree to practice a medically acceptable form of birth control.
* Intends to complete the study and willing to follow all study directions.

Exclusion Criteria:

* Allergies/sensitivity to skincare products or the test product ingredients
* Has a light or photosensitivity disorder or another medical condition that could increase risk to the subject or confuse the study results.
* Is taking medication that may cause skin sensitivity to light
* Has been using a product or medication that the study investigator determines will increase health risk to the subject or confuse the study results
* Has a facial skin condition (e.g. rosacea, acne, eczema, etc.) that could increase health risk to the subject or confuse the study results.
* Has skin cancer or a history of skin cancer.
* Has an immune deficiency disorder, active hepatitis, or an autoimmune disease.
* Has an uncontrolled metabolic condition (e.g. diabetes, hypertension)
* Is pregnant, nursing, or planning to become pregnant.
* Plans to start or change a hormone replacement therapy during the study.
* Has participated in another study in the past 30 days or plans to during the study.
* Is an employee or relative of the Study Site, Investigator, or Sponsor.

Ages: 35 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2017-10-09 (Actual); Primary Completion 2018-01-12 (Actual); Study Completion 2018-04-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stuart Lessin, M.D., Principal Investigator — KGL Skin Study Center, LLC
Locations (1):
- KGL Skin Study Center, LLC, Broomall, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fitzpatrick RE. Laser resurfacing of rhytides. Dermatol Clin. 1997 Jul;15(3):431-47. doi: 10.1016/s0733-8635(05)70452-6. PMID 9189680
- [Background] McCullough JL, Kelly KM. Prevention and treatment of skin aging. Ann N Y Acad Sci. 2006 May;1067:323-31. doi: 10.1196/annals.1354.044. PMID 16804006
- [Background] Weiss RA, McDaniel DH, Geronemus RG. Review of nonablative photorejuvenation: reversal of the aging effects of the sun and environmental damage using laser and light sources. Semin Cutan Med Surg. 2003 Jun;22(2):93-106. doi: 10.1053/sder.2003.50008. PMID 12877228
- [Background] Kim JW. Clinical trial of nonthermal 633 nm Omnilux LED array for renewal of photoaging: clinical surface profile metric results. Korea Soc Las Med Surg. 2005; 9:69-76.
- [Background] Fitzpatrick RE, Goldman MP, Satur NM, Tope WD. Pulsed carbon dioxide laser resurfacing of photo-aged facial skin. Arch Dermatol. 1996 Apr;132(4):395-402. PMID 8629842
- [Background] Griffiths CE, Wang TS, Hamilton TA, Voorhees JJ, Ellis CN. A photonumeric scale for the assessment of cutaneous photodamage. Arch Dermatol. 1992 Mar;128(3):347-51. PMID 1550366

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: At Visit 1 (Screening), participants were enrolled in the study and randomized to the active cell or the sham cell (stratified by skin type). All participants received the same facial cleanser and moisturizer with SPF to use between Visit 1 and Visit 2, and then received the assigned test product (Active Mask or Sham Mask) at Visit 2 (Baseline).
Groups:
- Sham Cell: Sham Mask: A facial cleanser was used twice daily (morning and evening). In the morning after washing, the moisturizer with SPF was applied full-face. For the first 12 weeks of the study, the sham light therapy mask was used for 10 minutes in the evening after washing/drying the face. For the second 12 weeks of the study, mask usage was discontinued.
- Active Cell: Active Mask: A facial cleanser was used twice daily (morning and evening). In the morning after washing, the moisturizer with SPF was applied full-face. For the first 12 weeks of the study, the active light therapy mask was used for 10 minutes in the evening after washing/drying the face. For the second 12 weeks of the study, mask usage was discontinued.
Period: Before Treatment (Screening to Baseline)
Arm/Group | Sham Cell: Sham Mask | Active Cell: Active Mask
Started | 61 | 63
Completed | 60 | 59
Not Completed | 1 | 4
Not completed — Lost to Follow-up | 0 | 2
Not completed — Withdrawal by Subject | 1 | 2
Period: Treatment (Baseline to Week 12)
Arm/Group | Sham Cell: Sham Mask | Active Cell: Active Mask
Started | 60 | 59
Completed | 56 | 54
Not Completed | 4 | 5
Not completed — Withdrawal by Subject | 3 | 4
Not completed — Protocol Violation | 1 | 1
Period: Regression (Week 12 to Week 24)
Arm/Group | Sham Cell: Sham Mask | Active Cell: Active Mask
Started | 56 | 54
Completed | 55 | 52
Not Completed | 1 | 2
Not completed — Protocol Violation | 1 | 1
Not completed — Death | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sham Cell: Sham Mask | Active Cell: Active Mask | Total
Number analyzed (Participants) | 61 | 63 | 124
Age, Continuous [Mean (Standard Deviation); unit: Years] | 56.3 (8.02) | 56.6 (7.34) | 56.5 (7.65)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 61 | 63 | 124
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 60 | 62 | 122
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 15 | 18 | 33
  White | 45 | 45 | 90
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Fitzpatrick Skin Type [Count of Participants; unit: Participants] — Measure of skin type characteristics including sensitivity to burning/tanning. Ranges from I to VI, where I = white, very fair; red or blond hair; blue eyes; freckles; always burns easily, never tans. VI = Black; black hair, black eyes. Never burns, deeply pigmented.
  Participants
    I | 11 | 11 | 22
    II | 11 | 11 | 22
    III | 9 | 11 | 20
    IV | 10 | 11 | 21
    V | 10 | 9 | 19
    VI | 10 | 10 | 20
Skin Oiliness Level [Count of Participants; unit: Participants] — Self-perceived facial skin type in terms of oiliness level with answer choices of oily, dry, normal, or combination skin.
  Participants
    Oily | 2 | 4 | 6
    Dry | 9 | 13 | 22
    Normal | 23 | 17 | 40
    Combination | 27 | 29 | 56

OUTCOME MEASURES:

1. Primary Outcome: Global Wrinkling - Change From Baseline to Week 12, Averaged Expert Grader Scores
Description: 3 Expert Graders evaluated global wrinkling on a 1-9 scale, where 1 = mildest wrinkles to 9 = most severe wrinkles. The 3 Expert Grader scores were averaged for Baseline and for Week 12. Change from baseline was calculated as Baseline mean minus Week 12 mean so a positive score indicates improvement.
Time Frame: Baseline to Week 12
Population: Intent-to-treat population was used, including all subjects with data for this time point. Missing values were imputed by carrying forward the last observed post-baseline score. 5 subjects withdrew prior to baseline and there was no post-baseline data to carry forward for an additional 3 subjects.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Sham Cell: Sham Mask | Active Cell: Active Mask
Number analyzed (Participants) | 59 | 57
Units on a scale | 0.18 (0.328) | 0.30 (0.341)
Statistical Analysis 1: Comparison: Sham Cell: Sham Mask; Test type: Superiority — Superiority to baseline concluded if the lower bound of the 95% confidence interval for the mean difference is above 0.5; p < 0.001, t-test, 2 sided; Mean Difference (Net) = 0.18, 95% CI 2-sided [0.09 to 0.26], Standard Deviation 0.328
Statistical Analysis 2: Comparison: Active Cell: Active Mask; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.001, t-test, 2 sided; Mean Difference (Net) = 0.30, 95% CI 2-sided [0.21 to 0.39], Standard Deviation 0.341
Statistical Analysis 3: Comparison: Sham Cell: Sham Mask vs Active Cell: Active Mask; Test type: Other — The null hypothesis was that the change from baseline to Week 12 was equal for the active cell and the sham cell. The alternative hypothesis was that the mean change from Baseline was not equal between the two cells; p = 0.025, ANCOVA; With treatment and skin type group as factors and the corresponding averaged baseline score as a covariate; Mean Difference (Net) = 0.14, 95% CI 2-sided [0.02 to 0.25], Standard Error of Mean 0.060

2. Primary Outcome: Global Wrinkling - Change From Baseline to Week 12, Individual Expert Grader Scores - Expert Grader 1
Description: Each Expert Graders evaluated global wrinkling on a 1-9 scale, where 1 = mildest wrinkles to 9 = most severe wrinkles. Change from baseline was calculated as Baseline mean minus Week 12 mean so a positive score indicates improvement. Scores for Expert Grader 1 were calculated individually.
Time Frame: Baseline to Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale.
Arm/Group | Sham Cell: Sham Mask | Active Cell: Active Mask
Number analyzed (Participants) | 59 | 57
Units on a scale. | 0.20 (0.349) | 0.22 (0.328)
Statistical Analysis 1: Comparison: Sham Cell: Sham Mask; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.001, t-test, 2 sided; Mean Difference (Net) = 0.20, 95% CI 2-sided [0.11 to 0.29], Standard Deviation 0.349
Statistical Analysis 2: Comparison: Active Cell: Active Mask; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.001, t-test, 2 sided; Mean Difference (Net) = 0.22, 95% CI 2-sided [0.13 to 0.31], Standard Deviation 0.328
Statistical Analysis 3: Comparison: Sham Cell: Sham Mask vs Active Cell: Active Mask; Test type: Equivalence — [test comment as in outcome 1, analysis 3]; p = 0.540, ANCOVA; With treatment and skin type group as factors and the corresponding averaged baseline score as a covariate; Mean Difference (Net) = 0.04, 95% CI 2-sided [-0.09 to 0.16], Standard Error of Mean 0.062

3. Primary Outcome: Global Wrinkling - Change From Baseline to Week 12, Individual Expert Grader Scores - Expert Grader 2
Description: Each Expert Graders evaluated global wrinkling on a 1-9 scale, where 1 = mildest wrinkles to 9 = most severe wrinkles. Change from baseline was calculated as Baseline mean minus Week 12 mean so a positive score indicates improvement. Scores for Expert Grader 2 were calculated individually.
Time Frame: Baseline to Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale.
Arm/Group | Sham Cell: Sham Mask | Active Cell: Active Mask
Number analyzed (Participants) | 59 | 57
Units on a scale. | -0.03 (0.532) | 0.21 (0.500)
Statistical Analysis 1: Comparison: Sham Cell: Sham Mask; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.627, t-test, 2 sided; Mean Difference (Net) = -0.03, 95% CI 2-sided [-0.17 to 0.10], Standard Deviation 0.532
Statistical Analysis 2: Comparison: Active Cell: Active Mask; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.002, t-test, 2 sided; Mean Difference (Net) = 0.21, 95% CI 2-sided [0.08 to 0.34], Standard Deviation 0.500
Statistical Analysis 3: Comparison: Sham Cell: Sham Mask vs Active Cell: Active Mask; Test type: Equivalence — [test comment as in outcome 1, analysis 3]; p = 0.009, ANCOVA; With treatment and skin type group as factors and the corresponding averaged baseline score as a covariate; Mean Difference (Net) = 0.24, 95% CI 2-sided [0.06 to 0.42], Standard Error of Mean 0.092

4. Primary Outcome: Global Wrinkling - Change From Baseline to Week 12, Individual Expert Grader Scores - Expert Grader 3
Description: Each Expert Graders evaluated global wrinkling on a 1-9 scale, where 1 = mildest wrinkles to 9 = most severe wrinkles. Change from baseline was calculated as Baseline mean minus Week 12 mean so a positive score indicates improvement. Scores for Expert Grader 3 were calculated individually.
Time Frame: Baseline to Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale.
Arm/Group | Sham Cell: Sham Mask | Active Cell: Active Mask
Number analyzed (Participants) | 59 | 57
Units on a scale. | 0.36 (0.465) | 0.47 (0.578)
Statistical Analysis 1: Comparison: Sham Cell: Sham Mask; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.001, t-test, 2 sided; Mean Difference (Net) = 0.36, 95% CI 2-sided [0.23 to 0.48], Standard Deviation 0.465
Statistical Analysis 2: Comparison: Active Cell: Active Mask; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.001, t-test, 2 sided; Mean Difference (Net) = 0.47, 95% CI 2-sided [0.32 to 0.63], Standard Deviation 0.578
Statistical Analysis 3: Comparison: Sham Cell: Sham Mask vs Active Cell: Active Mask; Test type: Equivalence — [test comment as in outcome 1, analysis 3]; p = 0.224, ANCOVA; With treatment and skin type group as factors and the corresponding averaged baseline score as a covariate; Mean Difference (Net) = 0.11, 95% CI 2-sided [-0.07 to 0.30], Standard Error of Mean 0.094

5. Secondary Outcome: Global Wrinkling - Change From Baseline to Week 1
Description: 3 Expert Graders evaluated global wrinkling on a 1-9 scale, where 1 = mildest wrinkles to 9 = most severe wrinkles. The 3 Expert Grader scores were averaged for Baseline and for Week 1. Change from baseline was calculated as Baseline mean minus Week 1 mean so a positive score indicates improvement.
Time Frame: Baseline to Week 1
Population: Intent-to-treat population was used, including all subjects with data for this time point. The number analyzed may be less than the total due to subject withdrawal prior to this time point or missed visits/evaluations.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Sham Cell: Sham Mask | Active Cell: Active Mask
Number analyzed (Participants) | 59 | 57
Units on a scale | 0.03 (0.158) | 0.04 (0.157)

6. Secondary Outcome: Global Wrinkling - Change From Baseline to Week 4
Description: 3 Expert Graders evaluated global wrinkling on a 1-9 scale, where 1 = mildest wrinkles to 9 = most severe wrinkles. The 3 Expert Grader scores were averaged for Baseline and for Week 4. Change from baseline was calculated as Baseline mean minus Week 4 mean so a positive score indicates improvement.
Time Frame: Baseline to Week 4
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Sham Cell: Sham Mask | Active Cell: Active Mask
Number analyzed (Participants) | 56 | 56
Units on a scale | 0.09 (0.208) | 0.09 (0.198)

7. Secondary Outcome: Global Wrinkling - Change From Baseline to Week 24
Description: 3 Expert Graders evaluated global wrinkling on a 1-9 scale, where 1 = mildest wrinkles to 9 = most severe wrinkles. The 3 Expert Grader scores were averaged for Baseline and for Week 24. Change from baseline was calculated as Baseline mean minus Week 24 mean so a positive score indicates improvement.
Time Frame: Baseline to Week 24
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Sham Cell: Sham Mask | Active Cell: Active Mask
Number analyzed (Participants) | 55 | 52
Units on a scale | 0.24 (0.410) | 0.30 (0.378)

8. Secondary Outcome: Fine Lines - Change From Baseline to Week 1
Description: 3 Expert Graders evaluated fine lines on a 1-9 scale, where 1 = mildest fine lines to 9 = most severe fine lines. The 3 Expert Grader scores were averaged for Baseline and for Week 1. Change from baseline was calculated as Baseline mean minus Week 1 mean so a positive score indicates improvement.
Time Frame: 1 week
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Sham Cell: Sham Mask | Active Cell: Active Mask
Number analyzed (Participants) | 59 | 57
Units on a scale | 0.01 (0.132) | 0.05 (0.160)

9. Secondary Outcome: Fine Lines - Change From Baseline to Week 4
Description: 3 Expert Graders evaluated fine lines on a 1-9 scale, where 1 = mildest fine lines to 9 = most severe fine lines. The 3 Expert Grader scores were averaged for Baseline and for Week 4. Change from baseline was calculated as Baseline mean minus Week 4 mean so a positive score indicates improvement.
Time Frame: Baseline to Week 4
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Sham Cell: Sham Mask | Active Cell: Active Mask
Number analyzed (Participants) | 56 | 56
Units on a Scale | 0.08 (0.196) | 0.13 (0.205)

10. Secondary Outcome: Fine Lines - Change From Baseline to Week 12
Description: 3 Expert Graders evaluated fine lines on a 1-9 scale, where 1 = mildest fine lines to 9 = most severe fine lines. The 3 Expert Grader scores were averaged for Baseline and for Week 12. Change from baseline was calculated as Baseline mean minus Week 12 mean so a positive score indicates improvement.
Time Frame: Baseline to Week 12
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Sham Cell: Sham Mask | Active Cell: Active Mask
Number analyzed (Participants) | 56 | 54
Units on a Scale | 0.23 (0.309) | 0.32 (0.358)

11. Secondary Outcome: Fine Lines - Change From Baseline to Week 24
Description: 3 Expert Graders evaluated fine lines on a 1-9 scale, where 1 = mildest fine lines to 9 = most severe fine lines. The 3 Expert Grader scores were averaged for Baseline and for Week 24. Change from baseline was calculated as Baseline mean minus Week 24 mean so a positive score indicates improvement.
Time Frame: Baseline to Week 24
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Sham Cell: Sham Mask | Active Cell: Active Mask
Number analyzed (Participants) | 55 | 52
Units on a Scale | 0.28 (0.358) | 0.29 (0.349)

12. Secondary Outcome: Periorbital Wrinkles - Change From Baseline to Week 1
Description: 3 Expert Graders evaluated periorbital wrinkles on a 1-9 scale, where 1 = mildest wrinkles to 9 = most severe wrinkles. The 3 Expert Grader scores were averaged for Baseline and for Week 1. Change from baseline was calculated as Baseline mean minus Week 1 mean so a positive score indicates improvement.
Time Frame: Baseline to Week 1
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Sham Cell: Sham Mask | Active Cell: Active Mask
Number analyzed (Participants) | 59 | 57
Units on a Scale | 0.00 (0.176) | 0.01 (0.172)

13. Secondary Outcome: Periorbital Wrinkles - Change From Baseline to Week 4
Description: 3 Expert Graders evaluated periorbital wrinkles on a 1-9 scale, where 1 = mildest wrinkles to 9 = most severe wrinkles. The 3 Expert Grader scores were averaged for Baseline and for Week 4. Change from baseline was calculated as Baseline mean minus Week 4 mean so a positive score indicates improvement.
Time Frame: Baseline to Week 4
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Sham Cell: Sham Mask | Active Cell: Active Mask
Number analyzed (Participants) | 56 | 56
Units on a Scale | 0.10 (0.269) | 0.10 (0.246)

14. Secondary Outcome: Periorbital Wrinkles - Change From Baseline to Week 12
Description: 3 Expert Graders evaluated periorbital wrinkles on a 1-9 scale, where 1 = mildest wrinkles to 9 = most severe wrinkles. The 3 Expert Grader scores were averaged for Baseline and for Week 12. Change from baseline was calculated as Baseline mean minus Week 12 mean so a positive score indicates improvement.
Time Frame: Baseline to Week 12
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Sham Cell: Sham Mask | Active Cell: Active Mask
Number analyzed (Participants) | 56 | 64
Units on a Scale | 0.15 (0.355) | 0.30 (0.366)

15. Secondary Outcome: Periorbital Wrinkles - Change From Baseline to Week 24
Description: 3 Expert Graders evaluated periorbital wrinkles on a 1-9 scale, where 1 = mildest wrinkles to 9 = most severe wrinkles. The 3 Expert Grader scores were averaged for Baseline and for Week 24. Change from baseline was calculated as Baseline mean minus Week 24 mean so a positive score indicates improvement.
Time Frame: Baseline to Week 24
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Sham Cell: Sham Mask | Active Cell: Active Mask
Number analyzed (Participants) | 55 | 52
Units on a Scale | 0.22 (0.399) | 0.29 (0.401)

16. Secondary Outcome: Surface Roughness - Change From Baseline to Week 1
Description: 3 Expert Graders evaluated surface roughness on a 0-9 scale, where 0 = perfectly smooth to 9 = severe roughness (visible and tactile). The 3 Expert Grader scores were averaged for Baseline and for Week 1. Change from baseline was calculated as Baseline mean minus Week 1 mean so a positive score indicates improvement.
Time Frame: Baseline to Week 1
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Sham Cell: Sham Mask | Active Cell: Active Mask
Number analyzed (Participants) | 59 | 57
Units on a Scale | 0.35 (0.396) | 0.38 (0.386)

17. Secondary Outcome: Surface Roughness - Change From Baseline to Week 4
Description: 3 Expert Graders evaluated surface roughness on a 0-9 scale, where 0 = perfectly smooth to 9 = severe roughness (visible and tactile). The 3 Expert Grader scores were averaged for Baseline and for Week 4. Change from baseline was calculated as Baseline mean minus Week 4 mean so a positive score indicates improvement.
Time Frame: Baseline to Week 4
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Sham Cell: Sham Mask | Active Cell: Active Mask
Number analyzed (Participants) | 56 | 56
Units on a Scale | 0.79 (0.438) | 0.76 (0.520)

18. Secondary Outcome: Surface Roughness - Change From Baseline to Week 12
Description: 3 Expert Graders evaluated surface roughness on a 0-9 scale, where 0 = perfectly smooth to 9 = severe roughness (visible and tactile). The 3 Expert Grader scores were averaged for Baseline and for Week 12. Change from baseline was calculated as Baseline mean minus Week 12 mean so a positive score indicates improvement.
Time Frame: Baseline to Week 12
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Sham Cell: Sham Mask | Active Cell: Active Mask
Number analyzed (Participants) | 56 | 54
Units on a Scale | 0.94 (0.449) | 0.89 (0.576)

19. Secondary Outcome: Surface Roughness - Change From Baseline to Week 24
Description: 3 Expert Graders evaluated surface roughness on a 0-9 scale, where 0 = perfectly smooth to 9 = severe roughness (visible and tactile). The 3 Expert Grader scores were averaged for Baseline and for Week 24. Change from baseline was calculated as Baseline mean minus Week 24 mean so a positive score indicates improvement.
Time Frame: Week 24
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Sham Cell: Sham Mask | Active Cell: Active Mask
Number analyzed (Participants) | 55 | 52
Units on a Scale | 1.12 (0.549) | 0.95 (0.686)

20. Secondary Outcome: Uneven Skin Tone - Change From Baseline to Week 1
Description: 3 Expert Graders evaluated uneven skin tone on a 0-9 scale, where 0 = perfectly uniform/even skin tone to 9 = pronounced/severe uneven skin tone. The 3 Expert Grader scores were averaged for Baseline and for Week 1. Change from baseline was calculated as Baseline mean minus Week 1 mean so a positive score indicates improvement.
Time Frame: Baseline to Week 1
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Sham Cell: Sham Mask | Active Cell: Active Mask
Number analyzed (Participants) | 59 | 57
Units on a Scale | 0.04 (0.176) | 0.06 (0.119)

21. Secondary Outcome: Uneven Skin Tone - Change From Baseline to Week 4
Description: 3 Expert Graders evaluated uneven skin tone on a 0-9 scale, where 0 = perfectly uniform/even skin tone to 9 = pronounced/severe uneven skin tone. The 3 Expert Grader scores were averaged for Baseline and for Week 4. Change from baseline was calculated as Baseline mean minus Week 4 mean so a positive score indicates improvement.
Time Frame: Baseline to Week 4
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Sham Cell: Sham Mask | Active Cell: Active Mask
Number analyzed (Participants) | 56 | 56
Units on a Scale | 0.18 (0.282) | 0.23 (0.287)

22. Secondary Outcome: Uneven Skin Tone - Change From Baseline to Week 12
Description: 3 Expert Graders evaluated uneven skin tone on a 0-9 scale, where 0 = perfectly uniform/even skin tone to 9 = pronounced/severe uneven skin tone. The 3 Expert Grader scores were averaged for Baseline and for Week 12. Change from baseline was calculated as Baseline mean minus Week 12 mean so a positive score indicates improvement.
Time Frame: Baseline to Week 12
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Sham Cell: Sham Mask | Active Cell: Active Mask
Number analyzed (Participants) | 56 | 54
Units on a Scale | 0.36 (0.388) | 0.49 (0.487)

23. Secondary Outcome: Uneven Skin Tone - Change From Baseline to Week 24
Description: 3 Expert Graders evaluated uneven skin tone on a 0-9 scale, where 0 = perfectly uniform/even skin tone to 9 = pronounced/severe uneven skin tone. The 3 Expert Grader scores were averaged for Baseline and for Week 24. Change from baseline was calculated as Baseline mean minus Week 24 mean so a positive score indicates improvement.
Time Frame: Baseline to Week 24
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Sham Cell: Sham Mask | Active Cell: Active Mask
Number analyzed (Participants) | 55 | 52
Units on a Scale | 0.44 (0.378) | 0.52 (0.499)

24. Secondary Outcome: Mottled Hyperpigmentation - Change From Baseline to Week 1
Description: 3 Expert Graders evaluated mottled hyperpigmentation on a 0-9 scale, where 0 = none (perfectly even tone) to 9 = severe mottled hyperpigmentation. The 3 Expert Grader scores were averaged for Baseline and for Week 1. Change from baseline was calculated as Baseline mean minus Week 1 mean so a positive score indicates improvement.
Time Frame: Baseline to Week 1
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Sham Cell: Sham Mask | Active Cell: Active Mask
Number analyzed (Participants) | 59 | 57
Units on a Scale | -0.01 (0.166) | -0.02 (0.174)

25. Secondary Outcome: Mottled Hyperpigmentation - Change From Baseline to Week 4
Description: 3 Expert Graders evaluated mottled hyperpigmentation on a 0-9 scale, where 0 = none (perfectly even tone) to 9 = severe mottled hyperpigmentation. The 3 Expert Grader scores were averaged for Baseline and for Week 4. Change from baseline was calculated as Baseline mean minus Week 4 mean so a positive score indicates improvement.
Time Frame: Baseline to Week 4
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Sham Cell: Sham Mask | Active Cell: Active Mask
Number analyzed (Participants) | 56 | 56
Units on a Scale | 0.10 (0.313) | 0.15 (0.288)

26. Secondary Outcome: Mottled Hyperpigmentation - Change From Baseline to Week 12
Description: 3 Expert Graders evaluated mottled hyperpigmentation on a 0-9 scale, where 0 = none (perfectly even tone) to 9 = severe mottled hyperpigmentation. The 3 Expert Grader scores were averaged for Baseline and for Week 12. Change from baseline was calculated as Baseline mean minus Week 12 mean so a positive score indicates improvement.
Time Frame: Baseline to Week 12
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Sham Cell: Sham Mask | Active Cell: Active Mask
Number analyzed (Participants) | 56 | 54
Units on a Scale | 0.22 (0.456) | 0.39 (0.392)

27. Secondary Outcome: Mottled Hyperpigmentation - Change From Baseline to Week 24
Description: 3 Expert Graders evaluated mottled hyperpigmentation on a 0-9 scale, where 0 = none (perfectly even tone) to 9 = severe mottled hyperpigmentation. The 3 Expert Grader scores were averaged for Baseline and for Week 24. Change from baseline was calculated as Baseline mean minus Week 24 mean so a positive score indicates improvement.
Time Frame: Baseline to Week 24
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Sham Cell: Sham Mask | Active Cell: Active Mask
Number analyzed (Participants) | 55 | 52
Units on a Scale | 0.25 (0.467) | 0.31 (0.401)

28. Secondary Outcome: Sallowness/Yellowing - Change From Baseline to Week 1
Description: 3 Expert Graders evaluated sallowness/yellowing on a 0-9 scale, where 0 = none to 9 = severe. The 3 Expert Grader scores were averaged for Baseline and for Week 1. Change from baseline was calculated as Baseline mean minus Week 1 mean so a positive score indicates improvement.
Time Frame: Baseline to Week 1
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Sham Cell: Sham Mask | Active Cell: Active Mask
Number analyzed (Participants) | 59 | 57
Units on a Scale | -0.01 (0.276) | 0.01 (0.179)

29. Secondary Outcome: Sallowness/Yellowing - Change From Baseline to Week 4
Description: 3 Expert Graders evaluated sallowness/yellowing on a 0-9 scale, where 0 = none to 9 = severe. The 3 Expert Grader scores were averaged for Baseline and for Week 4. Change from baseline was calculated as Baseline mean minus Week 4 mean so a positive score indicates improvement.
Time Frame: Baseline to Week 4
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Sham Cell: Sham Mask | Active Cell: Active Mask
Number analyzed (Participants) | 56 | 56
Units on a Scale | 0.12 (0.247) | 0.12 (0.354)

30. Secondary Outcome: Sallowness/Yellowing - Change From Baseline to Week 12
Description: 3 Expert Graders evaluated sallowness/yellowing on a 0-9 scale, where 0 = none to 9 = severe. The 3 Expert Grader scores were averaged for Baseline and for Week 12. Change from baseline was calculated as Baseline mean minus Week 12 mean so a positive score indicates improvement.
Time Frame: Baseline to Week 12
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Sham Cell: Sham Mask | Active Cell: Active Mask
Number analyzed (Participants) | 56 | 54
Units on a Scale | 0.23 (0.390) | 0.33 (0.496)

31. Secondary Outcome: Sallowness/Yellowing - Change From Baseline to Week 24
Description: 3 Expert Graders evaluated sallowness/yellowing on a 0-9 scale, where 0 = none to 9 = severe. The 3 Expert Grader scores were averaged for Baseline and for Week 24. Change from baseline was calculated as Baseline mean minus Week 24 mean so a positive score indicates improvement.
Time Frame: Baseline to Week 24
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Sham Cell: Sham Mask | Active Cell: Active Mask
Number analyzed (Participants) | 55 | 52
Units on a Scale | 0.29 (0.445) | 0.32 (0.504)

32. Secondary Outcome: Lack of Radiance - Change From Baseline to Week 1
Description: 3 Expert Graders evaluated lack of radiance on a 0-9 scale, where 0 = none (extremely radiant) to 9 = severe dullness/matte appearance. The 3 Expert Grader scores were averaged for Baseline and for Week 1. Change from baseline was calculated as Baseline mean minus Week 1 mean so a positive score indicates improvement.
Time Frame: Baseline to Week 1
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Sham Cell: Sham Mask | Active Cell: Active Mask
Number analyzed (Participants) | 59 | 57
Units on a Scale | 0.07 (0.219) | 0.13 (0.258)

33. Secondary Outcome: Lack of Radiance - Change From Baseline to Week 4
Description: 3 Expert Graders evaluated lack of radiance on a 0-9 scale, where 0 = none (extremely radiant) to 9 = severe dullness/matte appearance. The 3 Expert Grader scores were averaged for Baseline and for Week 4. Change from baseline was calculated as Baseline mean minus Week 4 mean so a positive score indicates improvement.
Time Frame: Baseline to Week 4
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Sham Cell: Sham Mask | Active Cell: Active Mask
Number analyzed (Participants) | 56 | 56
Units on a Scale | 0.28 (0.357) | 0.37 (0.401)

34. Secondary Outcome: Lack of Radiance - Change From Baseline to Week 12
Description: 3 Expert Graders evaluated lack of radiance on a 0-9 scale, where 0 = none (extremely radiant) to 9 = severe dullness/matte appearance. The 3 Expert Grader scores were averaged for Baseline and for Week 12. Change from baseline was calculated as Baseline mean minus Week 12 mean so a positive score indicates improvement.
Time Frame: Baseline to Week 12
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Sham Cell: Sham Mask | Active Cell: Active Mask
Number analyzed (Participants) | 56 | 54
Units on a Scale | 0.41 (0.412) | 0.55 (0.493)

35. Secondary Outcome: Lack of Radiance - Change From Baseline to Week 24
Description: 3 Expert Graders evaluated lack of radiance on a 0-9 scale, where 0 = none (extremely radiant) to 9 = severe dullness/matte appearance. The 3 Expert Grader scores were averaged for Baseline and for Week 24. Change from baseline was calculated as Baseline mean minus Week 24 mean so a positive score indicates improvement.
Time Frame: Baseline to Week 24
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Sham Cell: Sham Mask | Active Cell: Active Mask
Number analyzed (Participants) | 55 | 52
Units on a Scale | 0.54 (0.454) | 0.59 (0.517)

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected from time of informed consent through subject's last study procedure (Week 24 unless terminated early). Serious adverse events (SAE) reported to the site were also reportable within 30 days of last procedure/visit and longer if considered study-related; there was no specific cut-off date for this reporting, but AEs/SAEs are shown in this posting for a collection period of approximately 6 months from last subject's visit (the time of this posting).
Description: The Investigator or a designee interviewed subjects for changes in health/medication at each visit, documenting any reported adverse events. The analysis population is all randomized subjects who used the investigational device (i.e. the subjects enrolled in the treatment period).
Arm/Group | Sham Cell: Sham Mask | Active Cell: Active Mask
All-Cause Mortality (participants affected / at risk) | 0/60 | 1/59
Serious Adverse Events (participants affected / at risk) | 0/60 | 1/59
Other Adverse Events (participants affected / at risk) | 4/60 | 5/59
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sham Cell: Sham Mask (N=60) | Active Cell: Active Mask (N=59)
Sudden Death (General disorders) | 0 (0) | 1 (1) — Subject died during the regression period. Event was classified as "not study-related."
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sham Cell: Sham Mask (N=60) | Active Cell: Active Mask (N=59)
Upper Respiratory Tract Infection (Infections and infestations) | 1 (1) | 5 (5)
Oral Herpes (Infections and infestations) | 3 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI must provide Sponsor 60 days to review any publication (unless expedited review requested); if it includes Sponsor's confidential info, written Sponsor approval is required. Sponsor may require another 60 days' delay to file a patent application.

DOCUMENTS (2):
  • Study Protocol (2017-09-26): https://cdn.clinicaltrials.gov/large-docs/43/NCT03312543/Prot_000.pdf
  • Statistical Analysis Plan (2018-05-23): https://cdn.clinicaltrials.gov/large-docs/43/NCT03312543/SAP_001.pdf